CLINICAL TRIAL: NCT05161806
Title: An Open-label, Single-arm, Multicenter Study in Patients With Neovascular Age-related Macular Degeneration to Evaluate the Safety of SOK583A1 (40 mg/mL), a Proposed Aflibercept Biosimilar Product, Provided in a Prefilled Syringe
Brief Title: Study of the Safety of Use of Intravitreal SOK583A1 Provided in a Prefilled Syringe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOK583A12304
Record Dates: First submitted 2021-12-15; First posted 2021-12-17 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: Open label study,; intravitreal injection,; biosimilar,; aflibercept,; PFS
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- SOK583A1 (40 mg/mL) (Experimental): participants received a single dose of 2 mg SOK583 in 0.05 mL (40 mg/mL) and completed the study
  Interventions: Drug: SOK583A1 (40 mg/mL); Device: Prefilled Syringe (PFS)

INTERVENTIONS:
Drug: SOK583A1 (40 mg/mL) — SOK583A1 provided in a Prefilled Syringe (PFS), which includes 2 mg aflibercept in 0.05 mL for IVT administration
  Other Names: aflibercept
Device: Prefilled Syringe (PFS) — Prefilled Syringe (PFS)

SUMMARY:
This was an open-label, single arm, multicenter, Phase IIIb study in subjects with (wet) nAMD, eligible for IVT aflibercept treatment.

DETAILED DESCRIPTION:
This was an open-label, single arm, multicenter, Phase IIIb study in subjects with nAMD, eligible for Intravitreal (IVT) aflibercept treatment.

Screening and Baseline could be performed on the same day.

Subjects with nAMD received a single dose of study treatment (2 mg SOK583 in 0.05 mL) in line with the Eylea US PI, which recommends a dose of 2 mg aflibercept (0.05 mL) administered by IVT injection. Only subjects already under IVT Eylea treatment and hence familiar with the IVT procedure were eligible for the study. Administration of the study treatment was embedded into their individual dosing schedule.

Demonstration of the safe use of the PFS containing SOK583A1 was based on the performance of at least 3 different ophthalmologist teams.

Follow-up visits were performed on-site on Day 8 (±2 days) and on Day 31 (+4 days - end of study visit). Subjects participated for 30 to 34 days in the study including Baseline and treatment on Day 1 (Screening and Baseline could be performed on the same day) and the last safety follow-up on Day 31 (a time window of plus 4 days was allowed for the last safety follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 50 years of age at baseline
* Subjects diagnosed with nAMD (uni- or bilateral)
* Subjects already under IVT Eylea treatment (last injection of the induction period or maintenance phase)

Exclusion Criteria:

* Active or recent (within 4 weeks) intraocular inflammation (grade trace or above) in the study eye at baseline, which is of clinical significance according to the investigator's judgment, such as active infections of the anterior segment; this includes conjunctivitis (except mild blepharitis), keratitis, scleritis, idiopathic or autoimmune associated uveitis or endophthalmitis
* Any uncontrolled ocular hypertension or glaucoma in the study eye (defined as intraocular pressure (IOP) ≥ 26 mmHg, despite treatment with anti-glaucomatous medication)
* History of a medical, ocular or non-ocular condition, that in the judgment of the investigator, would preclude a safe administration of investigational product
* Visual Acuity Score (VAS) worse than 20/200 on a Snellen chart, the generally accepted level of legal blindness
* Receipt of any systemic anti-VEGF within the last 6 months prior to enrollment
* Uncontrolled hypertension (defined as a systolic value ≥ 160 mmHg or diastolic value ≥ 100 mmHg at Screening)
* Subjects who do not comply with the local COVID-19 regulations of the study site

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Sandoz Investigational Site, Marietta, Georgia
  - Sandoz Investigational Site, Oak Forest, Illinois
  - Sandoz Investigational Site, Liverpool, New York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 3 study sites in the US. All 3 sites screened and treated participants.
Pre-assignment Details: All enrolled participants received a single dose of 2 mg SOK583 in 0.05 mL (40 mg/mL).
Period: Overall Study
Arm/Group | SOK583A1 (40 mg/mL)
Started | 30
Full Analysis Set (FAS) (FAS included all participants who received an injection of study treatment.) | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SOK583A1 (40 mg/mL)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.4 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events
Description: Number of participants with ocular treatment emergent adverse events were reported.
Time Frame: throughout the study, approximately 31 days
Population: Full analysis set (FAS): FAS included all participants who received an injection of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 (40 mg/mL)
Number analyzed (Participants) | 30
Participants | 2

2. Primary Outcome: Number of Participants With Non-ocular Treatment Emergent Adverse Events
Description: Number of participants with non ocular Treatment emergent adverse events were reported.
Time Frame: throughout the study, approximately 31 days
Population: Full analysis set (FAS): FAS included all participants who received an injection of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 (40 mg/mL)
Number analyzed (Participants) | 30
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study i.e. approximately 31 days
Description: Any signs or symptoms were collected throughout the study i.e. approximately 31 days
Arm/Group | SOK583A1 (40 mg/mL)
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOK583A1 (40 mg/mL) (N=30)
Foreign body sensation in eyes (Eye disorders) | 1
Intraocular pressure increased (Investigations) | 1
Hypertension (Vascular disorders) | 1
Ocular discomfort (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05161806/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT05161806/SAP_001.pdf